CLINICAL TRIAL: NCT01277822
Title: The 8 Weeks, Multicenter, Randomized, Double-blind, Clinical Study To Evaluate Efficacy Of Treatment With Losartan/Amlodipine 100/5 mg Combination Compared To Amlodipine 10 mg Monotherapy In Hypertensive Patients Who Are Not Appropriately Respond To Amlodipine 5 mg Monotherapy
Brief Title: Efficacy of Losartan + Amlodipine Compared to Amlodipine Alone in the Treatment of Uncontrolled High Blood Pressure (MK-0954F-399)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0954F-399
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Results first posted 2014-04-24 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
Keywords: Hypertension; Uncontrolled hypertension; High blood pressure; Uncontrolled high blood pressure; Untreated high blood pressure; Untreated hypertension; Essential hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — amlodipine-losartan drug combination; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Losartan/amlodipine Treatment Arm (Experimental): One combination tablet containing 100 mg losartan potassium and 5 mg amlodipine camsylate, orally, once daily, for 8 weeks. Participants will also receive 2 tablets of placebo for amlodipine 5mg orally, once daily for 8 weeks.
  Interventions: Drug: Losartan (+) amlodipine; Drug: Placebo to match amlodipine
- Amlodipine Treatment Arm (Active Comparator): 2 tablets each containing 5 mg amlodipine, orally, once daily, for 8 weeks. Participants will also receive 1 tablet of placebo for combination losartan/amlodipine orally, once daily for 8 weeks.
  Interventions: Drug: Placebo to match losartan/amlodipine tablets; Drug: Amlodipine camsylate

INTERVENTIONS:
Drug: Losartan (+) amlodipine — One tablet containing 100 mg losartan potassium and 5 mg amlodipine camsylate, orally, once daily, for 8 weeks.
  Other Names: COZAAR XQ™
  Arms: Losartan/amlodipine Treatment Arm
Drug: Placebo to match losartan/amlodipine tablets — One tablet containing placebo, orally, once daily, for 8 weeks.
  Arms: Amlodipine Treatment Arm
Drug: Amlodipine camsylate — 2 tablets each containing 5 mg amlodipine, orally, once daily, for 8 weeks.
  Arms: Amlodipine Treatment Arm
Drug: Placebo to match amlodipine — 2 tablets containing placebo, orally, once daily, for 8 weeks.
  Arms: Losartan/amlodipine Treatment Arm

SUMMARY:
This study will determine whether using losartan and amlodipine together will be non-inferior in lowering blood pressure than amlodipine alone.

ELIGIBILITY:
Inclusion criteria

* Participants with essential hypertension:

  * who are on single drug therapy
  * who are newly diagnosed and not yet taking any drug therapy, or have not had any drug therapy for at least 2 weeks prior to entering study
  * who have blood pressure readings of 90mmHg ≤ MSDBP < 110mmHg and 140mmHg ≤ MSSBP <180mmHg after 2 weeks wash-out for patients on single agent.
* Randomization (Visit 3)

  * After dosing of amlodipine 5mg for 6 weeks, blood pressure readings are:

    * 90mmHg ≤ MSDBP < 110mmHg and 140mmHg ≤ MSSBP < 180mmHg.

Exclusion criteria

* Participant with MSDBP ≥ 110mmHg or MSSBP ≥ 180mmHg.
* Participant currently taking ≥ 2 antihypertensive medications (note: fixed-dose combination medicine should be counted as the number of active ingredients).
* Participant with known secondary hypertension of any etiology.
* Participant with malignant hypertension or current evidence of impending or active malignant hypertension, including headache, papilledema, cardiac ischemia, or pulmonary congestion precipitated by elevated blood pressure.
* Participant with known intolerance, contraindication or hypersensitivity to any component of dihydropyridines, angiotensin II receptor blockers.
* Participant showing positive in pregnancy test, lactating woman, or woman who intends to get pregnant during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2011-05-30 (Actual); Primary Completion 2013-04-22 (Actual); Study Completion 2013-04-22 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Losartan/Amlodipine: One combination tablet containing 100 mg losartan potassium and 5 mg amlodipine camsylate, orally, once daily, for 8 weeks. Participants will also receive 2 tablets of placebo for amlodipine 5mg orally, once daily for 8 weeks.
- Amlodipine: 2 tablets each containing 5 mg amlodipine, orally, once daily, for 8 weeks. Participants will also receive 1 tablet of placebo for combination losartan/amlodipine orally, once daily for 8 weeks.
Period: Overall Study
Arm/Group | Losartan/Amlodipine | Amlodipine
Started | 168 | 166
Completed | 153 | 155
Not Completed | 15 | 11
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Contraindicated medication used | 2 | 1
Not completed — Participant moved | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan/Amlodipine | Amlodipine | Total
Number analyzed (Participants) | 168 | 166 | 334
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (10.5) | 51.8 (10.6) | 52.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 36 | 78
  Male | 126 | 130 | 256

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Diastolic Blood Pressure (MSDBP) at Week 8
Description: Diastolic blood pressure was assessed at baseline and after 8 weeks of treatment with the participant in a seated position using an auto sphygmomanometer. Three measurements were performed at 2-minute intervals and the average of the 3 values of was recorded.
Time Frame: Baseline and Week 8
Population: Full Analysis Set defined as all participants who were randomized, took at least 1 dose of study drug, and had blood pressure measurements at baseline and at least 1 post-randomization blood pressure measurement.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Losartan/Amlodipine | Amlodipine
Number analyzed (Participants) | 162 | 160
mmHg | -10.1 (7.6) | -8.8 (7.8)
Statistical Analysis 1: Comparison: Losartan/Amlodipine vs Amlodipine; Test type: Non-Inferiority or Equivalence — Non-inferiority margin was 3 mmHg as Korean Food and Drug Administration (KFDA) guidance; p = 0.1339, t-test, 2 sided; Last observed non-missing, post-baseline value was imputed for missing value. If no such value existed, the value was treated as missing in analysis; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-3.0 to 0.4], Standard Deviation 7.7

2. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure (MSDBP) at Week 4
Description: Diastolic blood pressure was assessed at baseline and after 4 weeks of treatment with the participant in a seated position using an auto sphygmomanometer. Three measurements were performed at 2-minute intervals and the average of the 3 values of was recorded.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Losartan/Amlodipine | Amlodipine
Number analyzed (Participants) | 156 | 156
mmHg | -9.3 (7.8) | -10.0 (7.9)
Statistical Analysis 1: Comparison: Losartan/Amlodipine vs Amlodipine; Test type: Superiority or Other; p = 0.4478, t-test, 2 sided — No imputation for missing data was performed

3. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (MSSBP) at Week 8
Description: Systolic blood pressure was assessed at baseline and after 8 weeks of treatment with the participant in a seated position using an auto sphygmomanometer. Three measurements were performed at 2-minute intervals and the average of the 3 values of was recorded.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Losartan/Amlodipine | Amlodipine
Number analyzed (Participants) | 162 | 160
mmHg | -15.0 (12.1) | -12.7 (10.7)
Statistical Analysis 1: Comparison: Losartan/Amlodipine vs Amlodipine; Test type: Superiority or Other; p = 0.0717, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (MSSBP) at Week 4
Description: Systolic blood pressure was assessed at baseline and after 4 weeks of treatment with the participant in a seated position using an auto sphygmomanometer. Three measurements were performed at 2-minute intervals and the average of the 3 values of was recorded.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Losartan/Amlodipine | Amlodipine
Number analyzed (Participants) | 156 | 156
mmHg | -12.5 (13.2) | -12.3 (10.9)
Statistical Analysis 1: Comparison: Losartan/Amlodipine vs Amlodipine; Test type: Superiority or Other; p = 0.8736, t-test, 2 sided; No imputation for missing data was performed

5. Secondary Outcome: Percentage of Participants Who Achieve Target Blood Pressure at Week 8
Description: Participants were evaluated at Week 8 to ascertain if target blood pressure had been obtained. Criteria for meeting target BP were: sitting diastolic BP (sitDBP) <90mmHg or sitting systolic BP (sitSBP) <140mmHg) or sitDBP change more than 10mmHg from baseline or sitSBP change more than 20mmHg from baseline.
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Losartan/Amlodipine | Amlodipine
Number analyzed (Participants) | 162 | 160
Percentage of Participants | 63.0 | 58.8
Statistical Analysis 1: Comparison: Losartan/Amlodipine vs Amlodipine; Test type: Superiority or Other; p = 0.2508, Chi-squared — No imputation for missing data was performed

6. Secondary Outcome: Percentage of Participants Who Achieve Target Blood Pressure at Week 4
Description: Participants were evaluated at Week 4 to ascertain if target blood pressure had been obtained. Criteria for meeting target BP were: sitting diastolic BP (sitDBP) <90mmHg or sitting systolic BP (sitSBP) <140mmHg) or sitDBP change more than 10mmHg from baseline or sitSBP change more than 20mmHg from baseline.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Losartan/Amlodipine | Amlodipine
Number analyzed (Participants) | 156 | 156
Percentage of Participants | 55.1 | 61.5
Statistical Analysis 1: Comparison: Losartan/Amlodipine vs Amlodipine; Test type: Superiority or Other; p = 0.2508, Chi-squared — No imputation for missing data was performed

7. Secondary Outcome: Percentage of Participants Who Had Peripheral Edema During the Study
Description: A pitting assessment of edema on both legs was performed at baseline and throughout the study. Participants were assessed in a seated position with both feet extended and the right ankle in a neutral dorsiflexion position. The index finger was pressed firmly over the bony prominence approximately 3cm proximal to the midpoint of the medial malleolus of the right ankle and will be held for three seconds. Presence of a residual indentation in the area after releasing pressure on the index finger was considered positive for pitting edema.
Time Frame: up to 8 weeks
Population: Safety Set defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Losartan/Amlodipine | Amlodipine
Number analyzed (Participants) | 168 | 166
Percentage of Participants | 6.5 | 5.4
Statistical Analysis 1: Comparison: Losartan/Amlodipine vs Amlodipine; Test type: Superiority or Other; p = 0.6646, Chi-squared

8. Secondary Outcome: Change From Baseline in Ankle Circumference at Week 8
Description: Each ankle was marked with a semi-permanent marker at approximately 3 cm proximal to the midpoint of the medial malleolus to aid consistency in the performance of the measurements. Ankle circumference was measured in both ankles at baseline and Week 8 using a tension controlled tape to minimize error.
Time Frame: Baseline and Week 8
Population: All participants who received at least 1 dose of study drug and had available data for ankle circumference.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Losartan/Amlodipine | Amlodipine
Number analyzed (Participants) | 163 | 161
mm
  Left Ankle | -0.6 (4.7) | -0.7 (4.4)
  Right Ankle | -0.5 (4.0) | -0.2 (4.2)
Statistical Analysis 1: Comparison: Losartan/Amlodipine vs Amlodipine; Test type: Superiority or Other; p = 0.7911, t-test, 2 sided — Left ankle: Last observed non-missing, post-baseline value was imputed for missing value. If no such value existed, the value was treated as missing in analysis
Statistical Analysis 2: Comparison: Losartan/Amlodipine vs Amlodipine; Test type: Superiority or Other; p = 0.5933, t-test, 2 sided — Right ankle: Last observed non-missing, post-baseline value was imputed for missing value. If no such value existed, the value was treated as missing in analysis

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: Safety Set defined as all participants who received at least 1 dose of study drug.
Groups:
- Losartan 100mg/Amlodipine 5mg: One combination tablet containing 100 mg losartan potassium and 5 mg amlodipine camsylate, orally, once daily, for 8 weeks. Participants will also receive 2 tablets of placebo for amlodipine 5mg orally, once daily for 8 weeks
- Amlodipine 10mg: 2 tablets each containing 5 mg amlodipine, orally, once daily, for 8 weeks. Participants will also receive 1 tablet of placebo for combination losartan/amlodipine orally, once daily for 8 weeks.
Arm/Group | Losartan 100mg/Amlodipine 5mg | Amlodipine 10mg
Serious Adverse Events (participants affected / at risk) | 6/168 | 5/166
Other Adverse Events (participants affected / at risk) | 6/168 | 11/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan 100mg/Amlodipine 5mg (N=168) | Amlodipine 10mg (N=166)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 1 (1)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
EXCORIATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (2)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (2)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan 100mg/Amlodipine 5mg (N=168) | Amlodipine 10mg (N=166)
HEADACHE (Nervous system disorders) | 6 (6) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No